CLINICAL TRIAL: NCT02027909
Title: A Comparison of Rate Response Performance in Pacemaker Patients With an Indication of Sinus Node Dysfunction.
Acronym: CRIPS
Status: Completed | Type: Observational
Sponsor: Arun Rao (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Arun Rao, Arun Rao, MD. FACC, Wellmont CVA Heart Institute
Organization: Wellmont CVA Heart Institute (Other)
Other Study IDs: CRIPS
Record Dates: First submitted 2013-12-31; First posted 2014-01-06 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Sinus Node Dysfunction
Keywords: Sinus Node Dysfunction
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Therapy group one: Lower rate of 60 bpm and out of the box rate response settings of an ADL Rate of 95 bpm and rate profile optimization on with the only change being adjusting the activity threshold from med/low to low.
  Interventions: Device: Reprogramming dual chamber pacemaker
- Therapy group two: Rate response programming will be determined by an exercise test consisting of a 2 minute hall walk will be performed at the 2 week follow up and set points will be manually adjusted to achieve an ADL rate of 95 bpm. Rate Profile Optimization will be turned off. Activity threshold is programmed to low.
  Interventions: Device: Reprogramming dual chamber pacemaker
- Therapy group three: Lower rate of 60 bpm and the ADL rate based upon 220- age x 55%. Activity threshold is programmed to low. Rate Profile Optimization will be turned ON.
  Interventions: Device: Reprogramming dual chamber pacemaker

INTERVENTIONS:
Device: Reprogramming dual chamber pacemaker — Reprogramming rate response feature in the Medtronic pacemaker to each arm with crossover
  Other Names: Medtronic dual chamber pacemaker

SUMMARY:
Providing ideal rate response to patients should improve their quality of life and ability to execute activities of daily living.

Medtronic pacemakers provide rate response pacing by utilizing dual zone programming to specify an "activities of daily living" (ADL) response rate and an "exertion" response rate. There is much data to support the target heart rate for an exercise response but the data to support the programming of the ADL rate is lacking.

DETAILED DESCRIPTION:
Medtronic pacemakers provide rate response pacing by utilizing dual zone programming to specify an "activities of daily living" (ADL) response rate and an "exertion" response rate. There is much data to support the target heart rate for an exercise response but the data to support the programming of the ADL rate is lacking.

Unpublished Holter data from our center indicates that the ADL rate for most patients in our practice is between 50-70bpm rather than 95bpm. Moreover, this increased ADL rate may impact diastolic filling times and adversely impact cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension
* Sinus node dysfunction
* New implantation of a dual chamber pacemaker due to symptomatic sinus dysfunction or chronotropic incompetence defined as exercise heart rate less than 100 beats per minute

Exclusion Criteria:

* Second or Third degree AV block
* Age less than 60 or greater than 95 years
* EF less than 45%
* Patients that are not ambulatory
* Persistent atrial fibrillation (atrial fibrillation lasting greater than 7 days)
* Permanent atrial fibrillation (atrial fibrillation lasting great than 1 year)

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New implantation of a dual chamber pacemaker due to symptomatic sinus dysfunction or chronotropic incompetence defined as exercise heart rate less than 100 beats per minute
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
symptom improvement | study duration of 9 mths
  Patient report symptoms by clinician interview and patient symptom questionnaire

SECONDARY OUTCOMES:
improvement seen on device interrogations and reported improvement of symptoms | study duration of 9 mths
  Two minute hall walk distance Heart rate histograms and sensor indicated rate profile obtained from device interrogation Patient reported symptoms Patient symptom questionnaire Quality of life as measured by SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rao, MD, Principal Investigator — Wellmont CVA Heart Institute
Locations (1):
- Wellmont CVA Heart Institute, Kingsport, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau CP, Leung SK. Clinical usefulness of rate adaptive pacing systems: what should we assess? Pacing Clin Electrophysiol. 1994 Dec;17(12 Pt 1):2233-5. doi: 10.1111/j.1540-8159.1994.tb02370.x. No abstract available. PMID 7885929
- [Background] Lau CP, Tai YT, Leung WH, Wong CK, Lee P, Chung FL. Rate adaptive pacing in sick sinus syndrome: effects of pacing modes and intrinsic conduction on physiological responses, arrhythmias, symptomatology and quality of life. Eur Heart J. 1994 Nov;15(11):1445-55. doi: 10.1093/oxfordjournals.eurheartj.a060413. PMID 7835358
- [Background] Oto MA, Muderrisoglu H, Ozin MB, Korkmaz ME, Karamehmetoglu A, Oram A, Oram E, Ugurlu S. Quality of life in patients with rate responsive pacemakers: a randomized, cross-over study. Pacing Clin Electrophysiol. 1991 May;14(5 Pt 1):800-6. doi: 10.1111/j.1540-8159.1991.tb04110.x. PMID 1712957